CLINICAL TRIAL: NCT02294227
Title: A Phase III, Randomized, Double-blind, Placebo-controlled Multicenter Study of Subcutaneous Secukinumab (150 mg) in Pre-filled Syringe, With or Without Loading Regimen, to Demonstrate Efficacy, Safety and Tolerability up to 2 Years in Patients With Active Psoriatic Arthritis (FUTURE 4)
Brief Title: 16-week Efficacy and 2-year Safety, Tolerability and Efficacy of Secukinumab in Participants With Active Psoriatic Arthritis
Acronym: FUTURE 4
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CAIN457F2336; 2014-003849-10 (EudraCT Number)
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Results first posted 2019-07-02 (Actual); Last update posted 2019-07-02 (Actual); Status verified 2019-06

CONDITIONS: Arthritis, Psoriatic
Keywords: AIN457; psoriatic arthritis; chronic inflammatory disease; loading regimen; secukinumab; self-injection
MeSH Terms: conditions — Arthritis, Psoriatic | interventions — secukinumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (3):
- Secukinumab 150 mg (Experimental): Secukinumab 150 mg s.c. with loading: Secukinumab 150 mg at Baseline, Weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4. After primary outcome evaluation, approval and implementation of Amendment 2 Secukinumab dose may have been escalated to 300 mg as judged appropriate by the investigator
  Interventions: Biological: Secukinumab
- Secukinumab 150 mg No load (Experimental): Secukinumab 150 mg s.c. without loading: Secukinumab 150 mg at baseline, followed by dosing every four weeks starting at Week 4, with Placebo at Weeks 1, 2 and 3. After primary outcome evaluation, approval and implementation of Amendment 2 Secukinumab dose may have been escalated to 300 mg as judged appropriate by the investigator
  Interventions: Biological: Secukinumab
- Placebo (Placebo Comparator): Placebo to Secukinumab at Baseline, Weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4 until Week 16/24, depending on patients responder status. From Week 16/24, patients were switched to Secukinumab 150 mg every four weeks. After primary outcome evaluation, approval and implementation of Amendment 2 Secukinumab dose may have been escalated to 300 mg as judged appropriate by the investigator
  Interventions: Other: Placebo

INTERVENTIONS:
Biological: Secukinumab — Secukinumab 150 mg (1 mL liquid formulation) in pre-filled syringes were supplied by Novartis. Each secukinumab 300 mg dose was given as two sc injections of secukinumab 150 mg.
  Arms: Secukinumab 150 mg; Secukinumab 150 mg No load
Other: Placebo — Placebo to secukinumab was also available in 1.0 mL liquid formulation in prefilled syringe to match the active drug.
  Arms: Placebo

SUMMARY:
The purpose of this study was to provide 16-week efficacy, safety and tolerability data versus placebo to support the use of secukinumab 150 mg by subcutaneous (s.c.) self-administration with or without a loading regimen and maintenance dosing using pre-filled syringe (PFS) and to assess efficacy, safety and tolerability up to 2 years in subjects with active PsA despite current or previous NSAID or DMARD therapy

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of Psoriatic Arthritis (PsA) classified by ClASsification criteria for Psoriatic ARthritis (CASPAR) criteria.
* Rheumatoid factor and anti-cyclic citrullinated peptide (CCP) antibodies negative.
* Diagnosis of active plaque psoriasis or nail changes consistent with psoriasis.
* Inadequate control of symptoms with NSAID.
* Other protocol-defined inclusion criteria do apply.

Exclusion Criteria:

* Chest X-ray or chest magnetic resonance imaging (MRI) with evidence of ongoing infectious or malignant process.
* Subjects taking high potency opioid analgesics.
* Previous exposure to secukinumab or other biologic drug directly targeting interleukin-17 (IL-17) or IL-17 receptor.
* Ongoing use of prohibited psoriasis treatments / medications.
* Subjects who have ever received biologic immunomodulating agents except for those targeting TNFα.
* Previous treatment with any cell-depleting therapies.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 341 (Actual)
Dates: Start 2015-05-29 (Actual); Primary Completion 2016-02-16 (Actual); Study Completion 2017-12-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (58):
- United States (18):
  - Novartis Investigative Site, Mesa, Arizona
  - Novartis Investigative Site, Upland, California
  - Novartis Investigative Site, Denver, Colorado
  - Novartis Investigative Site, Palm Harbor, Florida
  - Novartis Investigative Site, Sarasota, Florida
  - Novartis Investigative Site, Peoria, Illinois
  - Novartis Investigative Site, Shreveport, Louisiana
  - Novartis Investigative Site, Saint Clair Shores, Michigan
  - Novartis Investigative Site, St Louis, Missouri
  - Novartis Investigative Site, Lincoln, Nebraska
  - Novartis Investigative Site, Albany, New York
  - Novartis Investigative Site, Oklahoma City, Oklahoma
  - Novartis Investigative Site, Duncansville, Pennsylvania
  - Novartis Investigative Site, Charleston, South Carolina
  - Novartis Investigative Site, Greenville, South Carolina
  - Novartis Investigative Site, Mesquite, Texas
  - Novartis Investigative Site, Burlington, Vermont
  - Novartis Investigative Site, Seattle, Washington
- Australia (4):
  - Novartis Investigative Site, Kogarah, New South Wales
  - Novartis Investigative Site, Maroochydore, Queensland
  - Novartis Investigative Site, Hobart, Tasmania
  - Novartis Investigative Site, Malvern East, Victoria
- Belgium (3):
  - Novartis Investigative Site, Aalst
  - Novartis Investigative Site, Brussels
  - Novartis Investigative Site, Yvoir
- Bulgaria (2):
  - Novartis Investigative Site, Plovdiv
  - Novartis Investigative Site, Sofia
- Canada (4):
  - Novartis Investigative Site, Victoria, British Columbia
  - Novartis Investigative Site, Winnipeg, Manitoba
  - Novartis Investigative Site, Pointe-Claire, Quebec
  - Novartis Investigative Site, Trois-Rivières, Quebec
- Czechia (4):
  - Novartis Investigative Site, Bruntál, Czech Republic
  - Novartis Investigative Site, Hlučín, Czech Republic
  - Novartis Investigative Site, Prague, Czech Republic
  - Novartis Investigative Site, Uherské Hradiště, Czech Republic
- France (2):
  - Novartis Investigative Site, Le Mans
  - Novartis Investigative Site, Montpellier
- Germany (7):
  - Novartis Investigative Site, Erlangen
  - Novartis Investigative Site, Frankfurt am Main
  - Novartis Investigative Site, Göttingen
  - Novartis Investigative Site, Hamburg
  - Novartis Investigative Site, Herne
  - Novartis Investigative Site, Magdeburg
  - Novartis Investigative Site, Nienburg
- Italy (3):
  - Novartis Investigative Site, Rozzano, MI
  - Novartis Investigative Site, Verona, VR
  - Novartis Investigative Site, Bologna
- Poland (5):
  - Novartis Investigative Site, Bialystok
  - Novartis Investigative Site, Dopiewo
  - Novartis Investigative Site, Elblag
  - Novartis Investigative Site, Lodz
  - Novartis Investigative Site, Poznan
- Russia (4):
  - Novartis Investigative Site, Petrozavodsk
  - Novartis Investigative Site, Saint Petersburg
  - Novartis Investigative Site, Yaroslavl
  - Novartis Investigative Site, Yekaterinburg
- Novartis Investigative Site, Stockholm, Sweden
- Novartis Investigative Site, Leytonstone, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com

REFERENCES:
- [Derived] Mease PJ, Warren RB, Nash P, Grouin JM, Lyris N, Willems D, Taieb V, Eells J, McInnes IB. Comparative Effectiveness of Bimekizumab and Secukinumab in Patients with Psoriatic Arthritis at 52 Weeks Using a Matching-Adjusted Indirect Comparison. Rheumatol Ther. 2024 Jun;11(3):817-828. doi: 10.1007/s40744-024-00652-7. Epub 2024 Mar 6. PMID 38446397
- [Derived] Pournara E, Kormaksson M, Nash P, Ritchlin CT, Kirkham BW, Ligozio G, Pricop L, Ogdie A, Coates LC, Schett G, McInnes IB. Clinically relevant patient clusters identified by machine learning from the clinical development programme of secukinumab in psoriatic arthritis. RMD Open. 2021 Nov;7(3):e001845. doi: 10.1136/rmdopen-2021-001845. PMID 34795065
- [Derived] Kivitz AJ, Nash P, Tahir H, Everding A, Mann H, Kaszuba A, Pellet P, Widmer A, Pricop L, Abrams K. Efficacy and Safety of Subcutaneous Secukinumab 150 mg with or Without Loading Regimen in Psoriatic Arthritis: Results from the FUTURE 4 Study. Rheumatol Ther. 2019 Sep;6(3):393-407. doi: 10.1007/s40744-019-0163-5. Epub 2019 Jun 21. PMID 31228101
- See also: Introduction to clinical trials conducted by Novartis and to results of completed studies, with the aim of increasing the transparency of Novartis clinical research and making publicly available objective scientific information in a standardised format. — http://www.novartisclinicaltrials.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: There were 341 patients originally randomized to one of 2 trearment groups. Seven placebo patients discontinued before week 16 and therefore not switched to treatment. Only 334 patients received secukinumab treatment.
Pre-assignment Details: Patients were randomized 1:1:1.
Period: Overall Study
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo
Started | 114 | 113 | 114
Completed (Completed Week 104) | 89 | 88 | 95
Not Completed | 25 | 25 | 19
Not completed — Death | 0 | 0 | 1
Not completed — Subject/Guardian Decision | 6 | 3 | 7
Not completed — Physician Decision | 1 | 2 | 1
Not completed — Lost to Follow-up | 1 | 0 | 0
Not completed — Lack of Efficacy | 11 | 12 | 8
Not completed — Adverse Event | 6 | 8 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo | Total
Number analyzed (Participants) | 114 | 113 | 107 | 334
Age, Continuous [Mean (Standard Deviation); unit: Years] | 48.3 (12.17) | 50.4 (11.78) | 48.5 (12.12) | 49.0 (12.03)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47 | 51 | 43 | 141
  Male | 67 | 62 | 64 | 193
Race/Ethnicity, Customized [Number; unit: Participants]
  Asian | 1 | 0 | 0 | 1
  White | 113 | 113 | 107 | 333

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With American College of Rheumatology 20 (ACR20) Response
Description: The ACR20 response is defined by at least 20% decrease in the swollen and tender joint count, and at least 20% improvement in 3 of the following 5 criteria:
  Health Assessment Questionnaire - Disability Index, pain score on a visual analog scale, patient global assessment of disease activity, physician global assessment of disease activity and acute phase reactant [either erythrocyte sedimentation rate (ESR) or high sensitivity C-reactive protein (hsCRP)]. ACR20 is used to assess the efficacy of secukinumab, with or without loading, versus placebo.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS): all subjects from the randomized set to whom study treatment has been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo
Number analyzed (Participants) | 114 | 113 | 114
Participants | 47 | 45 | 21
Statistical Analysis 1: Comparison: Secukinumab 150 mg No Load vs Placebo; Test type: Superiority; p = 0.0002, Chi-squared; Odds Ratio (OR) = 3.07, 95% CI 2-sided [1.66 to 5.66]
Statistical Analysis 2: Comparison: Secukinumab 150 mg vs Placebo; Test type: Superiority; p = 0.0003, Chi-squared, Corrected; Odds Ratio (OR) = 3.24, 95% CI 2-sided [1.76 to 5.97]

2. Secondary Outcome: Disease Activity Score (DAS-C28-CRP) Score Change From Baseline Using MMRM at Week 16
Description: DAS28-CRP score change from baseline using MMRM up to Week 16. DAS-CRP values range between 2.0 and 10. The higher the score, the higher the disease severity.
  n: Number of subjects with measures at both baseline and the corresponding post baseline visit.
Time Frame: week 16
Population: Full Analysis Set (FAS): all subjects from the randomized set to whom study treatment has been assigned.
Measure: Least Squares Mean (Standard Error); unit: scores
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo
Number analyzed (Participants) | 114 | 113 | 114
scores | -0.98 (0.106) | -0.84 (0.106) | -0.21 (0.107)

3. Secondary Outcome: Psoriatic Area and Severity Index 75 (PASI75)
Description: PASI is a measure of disease activity based on extent of the disease, severity of erythema, scaling and thickness in different body areas affected by psoriasis. PASI75 is an improvement in the PASI score of at least 75% compared to baseline. PASI75 is used to assess the efficacy of secukinumab, with or without loading, versus placebo.
  PASI75 response using non-responder imputation and rescue penalty up to Week 16
Time Frame: 16 weeks
Population: The psoriasis subset included all full analysis set (FAS) patients who had ≥3% of the body surface area (BSA) affected by psoriatic skin involvement at baseline.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo
Number analyzed (Participants) | 55 | 54 | 62
Participants | 29 [4.90 to 42.38] | 27 [4.14 to 35.19] | 5

4. Secondary Outcome: Short Form Health Survey Physical Component Score (SF-36-PCS)
Description: SF-36 is a 36 item questionnaire which measures Quality of Life across eight domains, which are both physically and emotionally based. Two overall summary scores, the Physical Component Summary (PCS) and Mental Component Summary (MCS) can be computed. In this study, SF-36 PCS is used to assess improvement from baseline of at least one dose of secukinumab versus placebo. The SF-36 is a validated instrument measuring health-related quality of life across multiple disease states. It has 36 questions with 8 subscale scores and 2 summary scores (1) physical component summary=physical functioning, role-physical, bodily pain, and general health. There is no total overall score; scoring is done for both subscores and summary scores. For subscores and summary scores, 0 =worst score (or quality of life) and 100=best score. Change from Baseline= post-Baseline - Baseline value.
Time Frame: 16 weeks
Population: Full Analysis Set (FAS): all subjects from the randomized set to whom study treatment has been assigned.
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Groups:
- Placebo Non-responder: Placebo to Secukinumab at Baseline, Weeks 1, 2 and 3, followed by dosing every four weeks starting at Week 4 until Week 16/24, depending on patients responder status. From Week 16/24, patients were switched to Secukinumab 150 mg every four weeks. After primary outcome evaluation, approval and implementation of Amendment 2 Secukinumab dose may have been escalated to 300 mg as judged appropriate by the investigator
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo Non-responder
Number analyzed (Participants) | 114 | 113 | 77
scores on a scale | 3.42 (0.5676) | 3.44 (0.5678) | 0.63 (0.586)

5. Secondary Outcome: Number of Participants With American College of Rheumatology 50 (ACR50)
Description: The ACR50 response is defined by at least 50% decrease in the swollen and tender joint count, and at least 50% improvement in 3 of the following 5 criteria: Health Assessment Questionnaire, pain score on a visual analog scale, patient global assessment of disease activity, physician global assessment of disease activity and acute phase reactant [either erythrocyte sedimentation rate (ESR) or high sensitivity C-reactive protein (hsCRP)].
  ACR50 is used to assess the efficacy of secukinumab, with or without loading, versus placebo.
  This table is the ACR50 response using non-responder imputation and rescue penalty up to Week 16
Time Frame: 16 weeks
Population: Full Analysis Set (FAS): all subjects from the randomized set to whom study treatment has been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo
Number analyzed (Participants) | 114 | 113 | 114
Participants | 26 | 19 | 7

6. Secondary Outcome: Number of Participants With American College of Rheumatology 20 (ACR20) Response
Description: The ACR20 response is defined by at least 20% decrease in the swollen and tender joint count, and at least 20% improvement in 3 of the following 5 criteria: Health Assessment Questionnaire - Diability Index, pain score on a visual analog scale, patient global assessment of disease activity, physician global assessment of disease activity and acute phase reactant [either erythrocyte sedimentation rate (ESR) or high sensitivity C-reactive protein (hsCRP)]. ACR20 is used to assess the efficacy of secukinumab, with or without loading, versus placebo
Time Frame: 4 weeks
Population: Full Analysis Set (FAS): all subjects from the randomized set to whom study treatment has been assigned.
Measure: Count of Participants; unit: Participants
Arm/Group | Secukinumab 150 mg | Secukinumab 150 mg No Load | Placebo
Number analyzed (Participants) | 114 | 113 | 114
Participants | 33 | 26 | 22

ADVERSE EVENTS:
Time Frame: Adverse Events (AEs) are collected from First Patient First Visit (FPFV) until Last Patient Last Visit (LPLV). All AEs reported in this record are from date of First Patient First Treatment until Last Patient Last Visit up to approximately week 112
Description: Safety analysis is based on actual dose received. Pts who escalated from 150mg to 300mg are also analyzed at escalated dose Any AIN457 150 mg (n = 334): 114 AIN150 Load + 113 AIN150 No Load + 107 PBO-AIN150 Any AIN457 (n = 334): 114 AIN150 Load + 113 AIN150 No Load + 107 PBO-AIN150 Any AIN457 300mg (n=136): 46 up-titrators from AIN150 load + 45 up-titrators from AIN150 No Load + 45 up-titrators from PBO - AIN300 Placebo (n=114): 114 patients were randomized to the placebo arm
Groups:
- Any AIN457 150 mg: Any AIN457 150 mg
- Any AIN457 300 mg: Any AIN457 300 mg
- Any AIN457: Any AIN457
- Placebo: Placebo
Arm/Group | Any AIN457 150 mg | Any AIN457 300 mg | Any AIN457 | Placebo
All-Cause Mortality (participants affected / at risk) | 1/334 | 1/136 | 2/334 | 1/114
Serious Adverse Events (participants affected / at risk) | 47/334 | 12/136 | 59/334 | 5/114
Other Adverse Events (participants affected / at risk) | 252/334 | 89/136 | 267/334 | 61/114
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=334) | Any AIN457 300 mg (N=136) | Any AIN457 (N=334) | Placebo (N=114)
Acute myocardial infarction (Cardiac disorders) | 1 | 0 | 1 | 0
Coronary artery disease (Cardiac disorders) | 1 | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 2 | 0 | 2 | 0
Myocardial ischaemia (Cardiac disorders) | 1 | 0 | 1 | 0
Goitre (Endocrine disorders) | 1 | 0 | 1 | 0
Abdominal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Colitis ulcerative (Gastrointestinal disorders) | 0 | 1 | 1 | 0
Crohn's disease (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Inguinal hernia (Gastrointestinal disorders) | 1 | 0 | 1 | 0
Pancreatitis acute (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Non-cardiac chest pain (General disorders) | 0 | 1 | 1 | 0
Biliary colic (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 1 | 0
Drug-induced liver injury (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Hepatitis alcoholic (Hepatobiliary disorders) | 1 | 0 | 1 | 0
Immunosuppression (Immune system disorders) | 0 | 1 | 1 | 0
Atypical pneumonia (Infections and infestations) | 0 | 1 | 1 | 0
Bacterial pyelonephritis (Infections and infestations) | 1 | 0 | 1 | 0
Campylobacter gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0 | 1 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 1 | 0
Hepatitis A (Infections and infestations) | 1 | 0 | 1 | 0
Influenza (Infections and infestations) | 1 | 0 | 1 | 0
Pilonidal cyst (Infections and infestations) | 0 | 0 | 0 | 1
Pyelonephritis (Infections and infestations) | 0 | 1 | 1 | 0
Sepsis (Infections and infestations) | 1 | 0 | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Urosepsis (Infections and infestations) | 1 | 0 | 1 | 0
Viral upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 0
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Laceration (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Rib fracture (Injury, poisoning and procedural complications) | 2 | 0 | 2 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 1 | 1 | 2 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Upper limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 0
Alanine aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Aspartate aminotransferase increased (Investigations) | 1 | 0 | 1 | 0
Hyponatraemia (Metabolism and nutrition disorders) | 1 | 0 | 1 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Arthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Cervical spinal stenosis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Joint range of motion decreased (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Loose body in joint (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Musculoskeletal chest pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 3 | 0 | 3 | 0
Polyarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0
Adrenal adenoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Chronic lymphocytic leukaemia (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Fibroma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 1 | 2 | 0
Papillary thyroid cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Parathyroid tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Squamous cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Undifferentiated sarcoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 1 | 0
Uterine leiomyoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Balance disorder (Nervous system disorders) | 1 | 0 | 1 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 1 | 0
Cervicogenic headache (Nervous system disorders) | 0 | 0 | 0 | 1
Facial paralysis (Nervous system disorders) | 1 | 0 | 1 | 0
Syncope (Nervous system disorders) | 2 | 0 | 2 | 0
Device dislocation (Product Issues) | 1 | 0 | 1 | 0
Device fastener issue (Product Issues) | 1 | 0 | 1 | 0
Disorientation (Psychiatric disorders) | 1 | 0 | 1 | 0
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 1 | 0
Ureteric compression (Renal and urinary disorders) | 0 | 1 | 1 | 0
Adenomyosis (Reproductive system and breast disorders) | 0 | 1 | 1 | 0
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 0
Nasal turbinate hypertrophy (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Skin ulcer (Skin and subcutaneous tissue disorders) | 0 | 1 | 1 | 0
Hypertensive crisis (Vascular disorders) | 1 | 0 | 1 | 0
Peripheral arterial occlusive disease (Vascular disorders) | 0 | 1 | 1 | 0
Raynaud's phenomenon (Vascular disorders) | 1 | 0 | 1 | 0
Thrombophlebitis (Vascular disorders) | 1 | 0 | 1 | 0
Varicose vein (Vascular disorders) | 1 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Any AIN457 150 mg (N=334) | Any AIN457 300 mg (N=136) | Any AIN457 (N=334) | Placebo (N=114)
Leukopenia (Blood and lymphatic system disorders) | 9 | 3 | 12 | 0
Ventricular extrasystoles (Cardiac disorders) | 3 | 3 | 6 | 0
Vertigo (Ear and labyrinth disorders) | 8 | 1 | 9 | 1
Abdominal pain (Gastrointestinal disorders) | 10 | 1 | 11 | 1
Diarrhoea (Gastrointestinal disorders) | 29 | 4 | 32 | 3
Dyspepsia (Gastrointestinal disorders) | 6 | 3 | 9 | 0
Nausea (Gastrointestinal disorders) | 19 | 2 | 21 | 6
Toothache (Gastrointestinal disorders) | 3 | 3 | 5 | 0
Vomiting (Gastrointestinal disorders) | 8 | 2 | 10 | 1
Fatigue (General disorders) | 13 | 3 | 16 | 2
Oedema peripheral (General disorders) | 5 | 2 | 7 | 1
Pyrexia (General disorders) | 11 | 1 | 12 | 1
Hepatic steatosis (Hepatobiliary disorders) | 6 | 2 | 8 | 0
Bronchitis (Infections and infestations) | 31 | 8 | 38 | 2
Cystitis (Infections and infestations) | 7 | 3 | 10 | 1
Furuncle (Infections and infestations) | 6 | 1 | 7 | 0
Gastroenteritis (Infections and infestations) | 15 | 5 | 19 | 3
Gastroenteritis viral (Infections and infestations) | 7 | 1 | 8 | 1
Gingivitis (Infections and infestations) | 6 | 1 | 7 | 2
Influenza (Infections and infestations) | 11 | 4 | 14 | 2
Laryngitis (Infections and infestations) | 5 | 3 | 8 | 1
Nasopharyngitis (Infections and infestations) | 86 | 21 | 96 | 16
Oral herpes (Infections and infestations) | 11 | 4 | 13 | 3
Pharyngitis (Infections and infestations) | 23 | 4 | 25 | 1
Pulpitis dental (Infections and infestations) | 8 | 2 | 10 | 0
Respiratory tract infection (Infections and infestations) | 10 | 2 | 11 | 2
Rhinitis (Infections and infestations) | 9 | 5 | 14 | 1
Sinusitis (Infections and infestations) | 29 | 11 | 34 | 1
Tonsillitis (Infections and infestations) | 10 | 6 | 14 | 0
Upper respiratory tract infection (Infections and infestations) | 48 | 11 | 55 | 6
Urinary tract infection (Infections and infestations) | 17 | 1 | 18 | 4
Viral infection (Infections and infestations) | 6 | 2 | 8 | 1
Viral upper respiratory tract infection (Infections and infestations) | 11 | 2 | 13 | 1
Contusion (Injury, poisoning and procedural complications) | 10 | 1 | 11 | 1
Fall (Injury, poisoning and procedural complications) | 11 | 2 | 13 | 1
Limb injury (Injury, poisoning and procedural complications) | 10 | 1 | 11 | 0
Alanine aminotransferase increased (Investigations) | 7 | 1 | 8 | 1
Hepatic enzyme increased (Investigations) | 6 | 2 | 8 | 0
Weight increased (Investigations) | 6 | 1 | 7 | 1
Dyslipidaemia (Metabolism and nutrition disorders) | 9 | 1 | 9 | 4
Hypercholesterolaemia (Metabolism and nutrition disorders) | 13 | 4 | 17 | 1
Hyperlipidaemia (Metabolism and nutrition disorders) | 5 | 2 | 7 | 0
Vitamin D deficiency (Metabolism and nutrition disorders) | 6 | 1 | 7 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 11 | 4 | 15 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 14 | 2 | 15 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 7 | 2 | 9 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7 | 1
Psoriatic arthropathy (Musculoskeletal and connective tissue disorders) | 21 | 12 | 28 | 5
Rotator cuff syndrome (Musculoskeletal and connective tissue disorders) | 5 | 2 | 7 | 0
Spinal pain (Musculoskeletal and connective tissue disorders) | 6 | 1 | 7 | 0
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 3
Dizziness (Nervous system disorders) | 5 | 0 | 5 | 3
Headache (Nervous system disorders) | 25 | 5 | 30 | 10
Migraine (Nervous system disorders) | 6 | 1 | 7 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 16 | 0 | 16 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 13 | 3 | 16 | 1
Eczema (Skin and subcutaneous tissue disorders) | 7 | 0 | 7 | 2
Pruritus (Skin and subcutaneous tissue disorders) | 6 | 2 | 8 | 1
Psoriasis (Skin and subcutaneous tissue disorders) | 7 | 5 | 12 | 1
Rash (Skin and subcutaneous tissue disorders) | 6 | 2 | 8 | 0
Hypertension (Vascular disorders) | 28 | 2 | 30 | 4

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (ie, data from all sites) in the clinical trial.